CLINICAL TRIAL: NCT01047540
Title: A Double-blind Randomized Placebo Controlled Dose-finding Trial to Investigate Different Doses of a New Antiviral Drug in Subjects With Genital HSV Type 2 Infection
Brief Title: Safety and Efficacy Study for a New Antiviral Drug to Treat Genital Herpes Type 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AIC316-01-II-01
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: HSV-2
MeSH Terms: interventions — pritelivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose regimen 1 (Experimental)
  Interventions: Drug: AIC316
- Dose regimen 2 (Experimental)
  Interventions: Drug: AIC316
- Dose regimen 3 (Experimental)
  Interventions: Drug: AIC316
- Dose regimen 4 (Experimental)
  Interventions: Drug: AIC316
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIC316 — Oral administration
  Other Names: pritelivir
  Arms: Dose regimen 1
Drug: AIC316 — Oral administration
  Other Names: pritelivir
  Arms: Dose regimen 2
Drug: AIC316 — Oral administration
  Other Names: pritelivir
  Arms: Dose regimen 3
Drug: AIC316 — Oral administration
  Other Names: pritelivir
  Arms: Dose regimen 4
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The aim of the study is to find out whether AIC316 is safe and efficacious for the prevention of reactivation of genital herpes

ELIGIBILITY:
Inclusion Criteria:

* Adult, Immunocompetent men and women in good health of any ethnic group
* History of recurrent episodes of genital herpes for at least 12 months
* Seropositive for Herpes Simplex Virus HSV Type 2
* Body Mass Index (BMI) between 18 and 35 kg/m2

Exclusion Criteria:

* Present episode of genital herpes
* Intake of systemic drug against HSV or any topical application against HSV within 7 days before randomization for the trial
* Intake of systemic corticosteroids, other immunomodulating agents or any investigational agent within 3 months before randomization for the trial
* Positive results in any of the virology tests for human immunodeficiency virus antibody (HIV-Ab), hepatitis C antibody (HCV-Ab), hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBc-Ab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cetero Research Miami Gardens, Miami, Florida
  - Indiana University School of Medicine, Office for Research, Indianapolis, Indiana
  - Westover Heights Clinic, Portland, Oregon
  - University of Texas Health Science Centre, Center for Clincial Studies, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Wald A, Corey L, Timmler B, Magaret A, Warren T, Tyring S, Johnston C, Kriesel J, Fife K, Galitz L, Stoelben S, Huang ML, Selke S, Stobernack HP, Ruebsamen-Schaeff H, Birkmann A. Helicase-primase inhibitor pritelivir for HSV-2 infection. N Engl J Med. 2014 Jan 16;370(3):201-10. doi: 10.1056/NEJMoa1301150. PMID 24428466

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Regimen 1: AIC316: Day 1 20 mg, Day 2-28 5 mg QD, Oral administration
- Dose Regimen 2: AIC316: Day 1 100 mg, Day 2-28 25 mg QD, Oral administration
- Dose Regimen 3: AIC316: Day 1 300 mg, Day 2-28 75 mg QD, Oral administration
- Dose Regimen 4: AIC316: 400 mg QWK, Oral administration
- Placebo: Matching placebo: Oral administration
Period: Overall Study
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo
Started | 34 | 32 | 29 | 31 | 30
Full Analysis Set | 33 | 32 | 29 | 31 | 30
Completed | 29 | 32 | 26 | 31 | 29
Not Completed | 5 | 0 | 3 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 29 | 31 | 30 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (12.56) | 38.8 (12.00) | 41.6 (12.47) | 42.0 (11.79) | 43.1 (10.81) | 40.5 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 20 | 20 | 21 | 104
  Male | 11 | 11 | 9 | 11 | 9 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 5 | 4 | 5 | 7 | 29
  White | 25 | 27 | 20 | 23 | 21 | 116
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 5 | 2 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of 4 Different Doses of AIC316 and Matching Placebo With Respect to the Suppression of Herpes Simplex Virus Replication (Shedding Rate)
Description: Subjects were assessed for shedding rate as the percentage of number of swab days with at least one swab positive for HSV DNA relative to the total number of days with analyzable swabs. Measurement was based on presence of HSV DNA measured on the material collected from swabs taken at the visits by the investigator and daily swabbing of the anogenital region by the patient during the treatment and post-treatment period.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: percentage of swab days
Groups:
- Dose Regimen 1: AIC316: Day 1 20 mg, Day 2-28, 5 mg QD, Oral administration
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo
Number analyzed (Participants) | 33 | 32 | 29 | 31 | 30
percentage of swab days | 21.2 (23.79) | 9.2 (12.61) | 2.0 (4.00) | 5.2 (6.50) | 16.5 (18.61)

ADVERSE EVENTS:
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32 | 0/29 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32 | 0/29 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 27/33 | 26/32 | 27/29 | 23/31 | 23/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Regimen 1 (N=33) | Dose Regimen 2 (N=32) | Dose Regimen 3 (N=29) | Dose Regimen 4 (N=31) | Placebo (N=30)
Gastrointestinal Disorder (Gastrointestinal disorders) | 17 | 13 | 17 | 15 | 12
Nausea (Gastrointestinal disorders) | 9 | 5 | 5 | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 5 | 4 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 4 | 4 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0
Nervous System Disorders (Nervous system disorders) | 13 | 15 | 14 | 16 | 12
Headache (Nervous system disorders) | 12 | 14 | 11 | 14 | 12
Dizziness (Nervous system disorders) | 3 | 1 | 5 | 2 | 1
Infections and Infestations (Infections and infestations) | 12 | 8 | 8 | 8 | 10
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2 | 1 | 3 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 1 | 0 | 3
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 10 | 9 | 7 | 6 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1 | 5
Pain in the Extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 2 | 3
General Disorders and Administration Site Conditions (General disorders) | 7 | 6 | 8 | 3 | 8
Fatigue (General disorders) | 4 | 2 | 5 | 3 | 5
Pyrexia (General disorders) | 1 | 1 | 3 | 1 | 0
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 7 | 4 | 7 | 5 | 8
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 2 | 2 | 4
Pruritus Genital (Reproductive system and breast disorders) | 1 | 0 | 2 | 1 | 3
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 6 | 7 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 4 | 3
Psychiatric Disorders (Psychiatric disorders) | 3 | 4 | 5 | 4 | 3
Insomnia (Psychiatric disorders) | 2 | 3 | 3 | 2 | 2
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 2 | 6 | 5 | 7 | 3
Investigations (Investigations) | 1 | 1 | 4 | 2 | 5
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 1 | 1 | 5 | 2 | 0
Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 2 | 1 | 3 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes